CLINICAL TRIAL: NCT05475730
Title: Tunnel Access for Ridge Augmentation Using Xenogenous Bone, Hyaluronic Acid and Acellular Dermal Matrix
Brief Title: Tunnel Access for Lateral Alveolar Ridge Augmentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: D'Albis Dental (Other)
Responsible Party: Principal Investigator, Giuseppe D'Albis, Principal Investigator, D'Albis Dental
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2022
Record Dates: First submitted 2022-01-15; First posted 2022-07-27 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Bone Loss; Implant Site Injury
MeSH Terms: conditions — Bone Diseases, Metabolic | interventions — Bone Regeneration

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bone regeneration (Experimental): Minimally invasive horizontal bone augmentation using hyaluronic acid, deproteinized bovine bone and dermal matrix.
  Interventions: Procedure: bone and soft tissue augmentation

INTERVENTIONS:
Procedure: bone and soft tissue augmentation — A vertical full-thickness incision in the mesial aspect of the defect ridge.Microsurgery instruments is subsequently use to carefully elevate the full thickness of the mucosa.
  Extreme caution must be exercised during these maneuvers to avoid tissue perforation and to maintain the integrity of the periosteum.An dermal matrix is place into the tunnel.A pouch is create between the bone and the membrane and the mixed bone chips and hyaluronic acid are inserted into the tunnel until the desirable ridge dimensions are obtained. Primary closure of the vertical incisions was achieved with single interrupted sutures.
  Other Names: Bone regeneration

SUMMARY:
Minimally invasive procedures with the tunnel technique have been suggested to decrease patient post-operative discomfort and morbidity in oral bone regeneration. In the ridge augmentation tunnel technique, crestal incision and the release of the connective tissue are avoided in order to enhance the blood supply of the flap. This approach preserves the blood circulation and does not damage the periosteum The purpose of this study is to evaluate the clinical outcome of a minimally invasive technique for maxillofacial horizontal bone augmentation .

performed by using a collagen dermal matrix, deproteinized bovine bone and hyaluronic acid.

Collagen matrix is inserted into a sub-periosteal tunnel using microsurgical instruments. Deproteinized bovine bone in a hyaluronic acid carrier are placed and inserted repeatedly into the pocket and absorbable suture is used to close the vertical incision.

DETAILED DESCRIPTION:
Tunnel bone regeneration achieves treatment objectives using the least invasive surgical approach.The goal is to increase patient satisfaction, decrease post-operative discomfort and morbidity.Preservation of the integrity of the periosteum is a determining factor in reducing postoperative pain and improving wound vascularization.

The present study value the clinical results of a subperiosteal minimally invasive ridge horizontal augmentation technique.

The technique includes the use of a laparoscopic approach to deliver hyaluronic acid,xenograft and a dermal matrix into a subperiosteal pouch.

ELIGIBILITY:
Inclusion Criteria:

* • Patients had to be healthy according to System of the American Society of Anesthesiology (ASA) and aged 18 years or older

  * No general medical condition representing a contraindication to implant therapy
  * minimum 2 missing teeth in the maxilla or mandible from the canine to the second molar
  * No periodontal disease (periodontal probing depth <4 mm) or treated periodontitis
  * Good oral hygiene (full mouth plaque index<25%)
  * Adequate control of inflammation (full mouth bleeding on probing<25%)

Exclusion Criteria:

* smoking of more than 15 cigarettes a day
* untreated periodontal disease
* pregnancy or breastfeeding at date of inclusion
* acute infections
* keratinized mucosal tissue less than 2 mm.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Augmented tissue volume | 7 month
  The edentulous ridge will be scanned with an intraoral scan 3 times. First time: Initial situation. Second time: 5 months after regeneration. Third time: After implant placement. Will be evaluate the 3 scan in a cad-cam software to evaluate the ridge three-dimensional changes.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe D'Albis, Study Director — D'Albis Dental
Locations (1):
- Giuseppe D'Albis, Mola di Bari, Bari, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kfir E, Kfir V, Eliav E, Kaluski E. Minimally invasive guided bone regeneration. J Oral Implantol. 2007;33(4):205-10. doi: 10.1563/1548-1336(2007)33[205:MIGBR]2.0.CO;2. PMID 17912961
- [Result] Karmon B, Tavelli L, Rasperini G. Tunnel Technique with a Subperiosteal Bag for Horizontal Ridge Augmentation. Int J Periodontics Restorative Dent. 2020 Mar/Apr;40(2):223-230. doi: 10.11607/prd.4508. PMID 32032406
- [Result] Rasperini G, Tavelli L, Barootchi S, Karmon B. Tunnel Technique with a Subperiosteal Bag for Ridge Augmentation: A Case Series. Int J Periodontics Restorative Dent. 2021 Sep-Oct;41(5):693-700. doi: 10.11607/prd.5136. PMID 34547072